CLINICAL TRIAL: NCT01169662
Title: Effects of Dietary Nitrate From Vegetable/Fruit Juice on Cerebral Blood Flow Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Prof. David Kennedy, Northumbria University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24AE1
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Cerebrovascular Circulation; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Vegetables; Fruit and Vegetable Juices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegetable/ Fruit juice (Active Comparator): 450ml active product, 45 ml no added sugar squash (for flavour)
  Interventions: Dietary Supplement: Vegetable/fruit juice
- Placebo juice (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo juice

INTERVENTIONS:
Dietary Supplement: Vegetable/fruit juice — 450ml active juice, 45ml no added sugar fruit squash (for flavour)
  Arms: Vegetable/ Fruit juice
Dietary Supplement: Placebo juice — 50 ml No Added Sugar fruit squash, 45 ml Pressed Apple Juice, 405ml with water.
  Arms: Placebo juice

SUMMARY:
Nitrate provides the body with an alternative source of Nitric Oxide which plays a large role in promoting blood flow and reducing blood pressure. Nitrate supplementation with vegetable/fruit juice has recently been shown to reduce blood pressure and reduce energy expenditure during low intensity exercise. Such findings combined with the previously known biological effects of nitric oxide would suggest that nitrate supplementation would also impact on blood flow. The aim of this study is to examine the effects of dietary nitrate supplementation via vegetable/fruit juice drink on cerebral (brain) blood flow (using Near Infrared Spectroscopy).

ELIGIBILITY:
Inclusion Criteria:

* healthy young (18-35 years) male and female adults, not vulnerable.

Exclusion Criteria:

* smoke or consume any tobacco products (even occasionally)
* not proficient in English
* pregnant (or are seeking to become)
* currently taking recreational, over the counter/prescription medication (excluding the contraceptive pill), and/or dietary/herbal supplements.
* any food allergies or sensitivities that are relevant to the study
* history of/current head trauma, learning difficulties, ADHD, dyslexia, migraines or any gastric problems.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline cerebral blood flow | From baseline to 2.5 hours post-dose
  Near infrared spectroscopy monitoring of cerebral blood flow in the frontal cortex during demanding tasks. Monitored from baseline, through 90 minutes of drink absorption and 60 minutes of cognitive task performance.
Change from baseline cognitive function | 90 minutes post-dose
  Performance of the cognitive demand battery (CDB), which assesses aspects of psychomotor speed, working memory and executive function. The CDB involves 6 repetitions of the following tasks: serial three subtractions (2 mins); serial seven subtractions (2 mins); Rapid Visual Information Processing (5 mins) and a subjective rating of mental fatigue
Change from baseline mood | 2.5 hours post-dose
  Bond-Lader visual analogue mood scales assessing the mood factors 'alert'; 'calm'; and 'content'

SECONDARY OUTCOMES:
Change from baseline blood pressure, heart rate and venous nitrate and nitrite levels | 2.5 hours post-dose
  Diastolic and systolic blood pressure and heart rate monitored after completion of cognitive tasks to assess peripheral blood flow effects. Plasma nitrate and nitrite levels assessed at 2.5 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

REFERENCES:
- [Derived] Wightman EL, Haskell-Ramsay CF, Thompson KG, Blackwell JR, Winyard PG, Forster J, Jones AM, Kennedy DO. Dietary nitrate modulates cerebral blood flow parameters and cognitive performance in humans: A double-blind, placebo-controlled, crossover investigation. Physiol Behav. 2015 Oct 1;149:149-58. doi: 10.1016/j.physbeh.2015.05.035. Epub 2015 May 31. PMID 26037632